CLINICAL TRIAL: NCT01643096
Title: The Effect of Thyme and Sumac on the Thermic Effect of Food and Comparison Between Warm and Cold Temperament People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 90-04-27-15366
Record Dates: First submitted 2012-07-15; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Effects of; Food, Allergic
Keywords: Zataria multiflora Boiss Sumac TEF temperament

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sumac (Other): Thermic effect of food of Sumac and comparison between hot and cold temperament people
  Interventions: Other: Sumac
- Zataria multiflora Boiss (Other): Thermic effect of food of Zataria multiflora Boiss and comparison between hot and cold temperament people
  Interventions: Other: Zataria multiflora Boiss

INTERVENTIONS:
Other: Zataria multiflora Boiss — Thermic effect of food of Zataria multiflora Boiss and comparison between hot and cold temperament people
  Other Names: Thyme
  Arms: Zataria multiflora Boiss
Other: Sumac — Thermic effect of food of Sumac and comparison between hot and cold temperament people
  Other Names: sumach
  Arms: sumac

SUMMARY:
The purpose of this study is to determine the effect of Zataria multiflora Boiss and Sumac on the thermic effect of food, activity of sympathetic - parasympathetic system: comparison between warm and cold temperament people.

DETAILED DESCRIPTION:
Human body needs to energy in order to preserve life.There are three forms of energy consumption at body, consumption at baseline or resting, consumption at energy expenditure for Thermic effect of food and energy is spent in physical activity.Also from the perspective of traditional medicine, cold and warm natured people are determined based on certain mental and physical protests.

There are different temperament not only in Traditional Iranian Medicine, but in traditional Chinese medicine, Indian, Greek, Arabic, Romanian, and there are European.As various factors on the basal metabolism and thermic effect of food , also are several factors such as age, sex, physical condition of the environment that have an impact on individual temperament.

Since the protests seem warm and cool temperament and factors affecting on their basal metabolic rate and thermogenesis so that food may explain the relationship between warm and cold temperament to mind is the basal metabolism; It seems those are hot temperament, their basal metabolic rate is higher BMR than normal and those who are cold temperament, have a lower BMR.

On the other hand seems that thermic effect of food in people who have hot temperament is higher than thermic effect of food in people who have cold temperament.

So that we need to use of two nutrient foods, in this way we consided the multiple criteria and then were selected sumac and thyme.

On the other hand, in order to study possible mechanisms affecting basal metabolism, thermogenesis of food, according to previous studies and also matches that there are between sympathetic - parasympathetic and thyroid function, with symptoms of cold and warm temperament there, checking of activity of these organs seems necessary.

Because to maintain basal metabolic rate is essential for human life, so that each factor in order to better understand these is helpful to human life.And the need for such study makes clear;Through this step help toward improving public health

ELIGIBILITY:
Inclusion criteria:

* Age 18 to 40 years
* Having to suffer any ill health and lack of attention to history and physical examination
* Willing to cooperate with the project

Exclusion Criteria:

* Catching any disease.
* Use of specific dietary patterns such as vegetarianism
* Having a BMI outside the normal range
* Use of any drugs or supplements in past month
* Allergic reaction to food allergy and non-prescription
* An unwillingness to cooperate in any of the stages of implementation

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
Thermic Effect of Food (TEF) | Change from baseline to 4 hours And repeated 1 week later
  kilocalorie(kcal) and by indirect calorimetery

SECONDARY OUTCOMES:
activity of sympathetic - parasympathetic system(Epinephrine, Norepinephrine, Cortisol) | Change from baseline to 4 hours And repeated 1 week later
  ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Ahmadreza Dorosty Motlagh, PhD, Principal Investigator — Tehran University of Medical Sciences, tehran, iran
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran